CLINICAL TRIAL: NCT05234216
Title: Comparison of a Comfort Scale and a Numerical Pain Scale on Opioid Consumption After Surgery: The COMFORT Randomized Trial
Brief Title: Comparison of a Comfort Scale and a Numerical Pain Scale on Opioid Consumption After Surgery
Acronym: COMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC20_8999_COMFORT; 2021-A02839-32 (Other: ANSM)
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Pain Management; Analgesia
Keywords: Comfort scale; Pain scale; numerical verbal scale; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Informed Consent; Surgical Procedures, Operative; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, interventional, randomized cluster study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comfort Group (Experimental): Centers evaluating patients after surgery requiring postoperative opioid treatment with an ICU comfort scale.
  Interventions: Other: Informed consent; Procedure: Surgery; Behavioral: Comfort scale; Other: Questionnaires
- Pain Group (Other): Centers evaluating patients, after surgery requiring postoperative opioid treatment, with a pain numerical verbal scale in the postoperative care service.
  Interventions: Other: Informed consent; Procedure: Surgery; Behavioral: Pain; Other: Questionnaires

INTERVENTIONS:
Other: Informed consent — the investigator will verify the inclusion criteria, the patient's understanding of the protocol and will obtain oral informed consent
Procedure: Surgery — The patient will undergo surgery in accordance with standard care
Behavioral: Comfort scale — The patient will be evaluated, in the post-operative care unit, with a comfort scale
  Arms: Comfort Group
Behavioral: Pain — The patient will be evaluated, in the post-operative care unit, with a pain scale
  Arms: Pain Group
Other: Questionnaires — Evaluation of the Experience of Local/General Anesthesia

SUMMARY:
The objective is to show that the use of therapeutic communication tools, in this case a comfort scale, a low cost and simple to implement method, can reduce pain and therefore the consumption of opioids in the postoperative care unit.

Our hypothesis is that the use of a comfort scale will lead to significant postoperative opioid sparing, and consequently to a decrease in the opioid-related side effects The aim of this study is to compare postoperative opioid consumption between patients whose pain is assessed by a numerical verbal scale and those assessed with a comfort scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient eligible for any surgery requiring postoperative opioid administration;
* Patient with a social security plan;
* French-speaking patient
* Free, informed and oral consent by the patient.

Exclusion Criteria:

* Woman claiming to be pregnant or breast feeding;
* Emergency surgery;
* Patients using preoperative opioids ;
* Opioid addiction;
* Patients unable to understand the assessment scales;
* Adults under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Opiate consumption in the post-operative care service | 1 day
  Opiate consumption in milligrams in the post-operative care service in morphine equivalent.

SECONDARY OUTCOMES:
Opioid consumption in the post-operative care service according to Ambulatory or conventional management | 1 day
  Opioid consumption in mg in the post-operative care service in morphine equivalent according to Ambulatory or conventional management
Opioid consumption in the post-operative care service according to the Risk related to surgery (minor / intermediate / major) | 1 day
  Opioid consumption in mg in the post-operative care service according to the Risk related to surgery (minor / intermediate / major)
Opioid consumption in the post-operative care service according to the Type of surgery | 1 day
  Opioid consumption in mg in the post-operative care service according to the Type of surgery
Determine if the use of a comfort scale in the post-operative care servic is associated with better postoperative analgesia | 1 day
  Number of postoperative pain episodes (NRS pain > 3) expressed in the post-operative care servic after extubation, at rest
Determine if the use of a comfort scale can reduce the time to achieve a Kremlin Bicetre score = 0, or a modified Aldrete score ≥ 9 or a Chung score ≥ 9 (for ambulatory) ; | 1 day
  Time from extubation to Kremlin Bicetre score = 0, or modified Aldrete score ≥ 9 or Chung score ≥ 9 (for ambulatory) ;
Determine whether the use of a comfort scale reduces postoperative nausea and vomiting; | 1 day
  Number of postoperative nausea and vomiting episodes in the post-operative care service, the use of anti-emetic treatment will be assessed ;
Determine whether the use of a comfort scale is associated with improved postoperative satisfaction. | 1 day
  Satisfaction questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic MEURET, Principal Investigator — Rennes University Hospital
Locations (29):
- France (28):
  - Chu Rennes - Pontchaillou, Rennes, CHU de Rennes
  - CHRU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CH Pierre Oudot, Bourgoin
  - HIA Clermont Tonnerre, Brest
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - CH Sud Francilien, Corbeil-Essonnes
  - CH Dax, Dax
  - GHM de Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - CHRU Lille - Hôpital Huriez, Lille
  - CH Saint Joseph Saint Luc, Lyon
  - Clinique du Parc, Lyon
  - Clinique Juge, Marseille
  - Clinique Jules Verne, Nantes
  - APHP - Hôpital Bichat, Paris
  - APHP - Hôpital Cochin, Paris
  - Polyclinique Saint Laurent de Rennes, Rennes
  - CH Saint-Brieuc, Saint-Brieuc
  - Centre Hospitalier Privé St Grégoire, Saint-Grégoire
  - Clinique Saint-Jean Cap Santé, Saint-Jean-de-Védas
  - CHRU Strasbourg - Hôpital Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - CHU Toulouse - Hôpital Riquet, Toulouse
  - CHRU Tours - Hôpital Bretonneau, Tours
  - CH Bretagne Atlantique, Vannes
- Hôpital Hôtel Dieu de France, Beirut, Lebanon

REFERENCES:
- [Derived] Fusco N, Meuret L, Bernard F, Musellec H, Martin L, Leonard M, Lasocki S, Gazeau T, Aubertin R, Blayac D, Leviel F, Danguy des Deserts M, Madi-Jebara S, Fessler J, Lecoeur S, Cirenei C, Menut R, Lebreton C, Bouvier S, Bonnet C, Maurice-Szamburski A, Cattenoz M, El Alami M, Brocas E, Aveline C, Gueguen L, Noll E, Gouel-Cheron A, Evrard O, Fontaine M, Nguyen YL, Ravry C, Boselli E, Laviolle B, Beloeil H; COMFORT Study Group and the French Society of Anesthesiologists (SFAR) Research Network. Effect of a comfort scale compared with a pain numerical rate scale on opioids consumption in postanaesthesia care unit: the COMFORT study. Br J Anaesth. 2024 Oct;133(4):839-845. doi: 10.1016/j.bja.2024.06.029. Epub 2024 Sep 7. PMID 39244480